CLINICAL TRIAL: NCT03594669
Title: Sensorimotor Training for Injury Prevention in Collegiate Soccer Players
Brief Title: Training for Injury Prevention in Collegiate Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Mississippi College (Unknown)
Responsible Party: Principal Investigator, Jennifer C. Reneker, Associate Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17-0232
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This study will be conducted as pilot of a one-arm intervention using,1) pre- and post-participation measures of sensorimotor control and 2) injury incidence rate over the sports-season directly after completion of the intervention compared to injury incidence rate of a historical control (the 2017 soccer season at Mississippi College). Participants will include men and women athletes on soccer teams from one Division II institution.
Masking Description: No masking will be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): When enrolled into the study, the participants will be asked to join a group in WhatsApp for purposes of the research study. The application will be used to: deliver reminders for each treatment session; deliver daily prompts for the home exercise program; and present a web-link to the home exercise program (HEP).
  Participants will receive physical therapist delivered multi-modal sensorimotor training interventions. The exercises delivered at each intervention will be delivered in a group format, using a circuit of exercises that each athlete will complete in a session. Subsequent sessions will build upon previous sessions to work the sensorimotor control system in progressively more challenging and sport-specific scenarios. This present study will complete 8 sessions over 4 weeks.
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Multi-modal sensorimotor training interventions, including vestibular, oculomotor, neuromotor, and postural control/ balance exercises.

SUMMARY:
The purpose of this research project is to evaluate the effectiveness of an injury prevention intervention for collegiate soccer players.

DETAILED DESCRIPTION:
The purpose of this research project is to evaluate the effectiveness of an injury prevention intervention for collegiate soccer players. The hypothesis is that measures of sensorimotor control will improve and injury incidence rate will decrease after participation in an intervention aimed at restoration/refinement of sensorimotor control. This study will be conducted as a 1-arm intervention with pre- and post-participation measurement of sensorimotor control and completion of an exercise intervention. Statistical analyses will be completed to determine within group change pre-to post-intervention and injury risk by comparing injury rate in 2018 to injury rate of a historical control.

ELIGIBILITY:
Inclusion Criteria:

* Male and female athletes on the soccer roster who are eligible to play in the fall 2018 season at Mississippi College

Exclusion Criteria:

* Any athlete who has a current diagnosis of concussion (i.e. a non-medically cleared concussion), lower-extremity musculoskeletal injury, or other medical diagnosis that will prevent the athlete from participation in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-08-11 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in clinical measures of sensorimotor control | Pre to post-treatment (1 month)
  Clinical examination tests

SECONDARY OUTCOMES:
Injury incidence rate | 1 year
  b) The incidence rate ratio of injury rates between a historical control (2017 soccer season) and the 2018 soccer-season from the participating college's soccer teams.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Reneker, PT, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No